CLINICAL TRIAL: NCT05069454
Title: Cohort Study to Measure COVID-19 Vaccine Effectiveness Among Health Workers in Azerbaijan
Brief Title: Study on COVID-19 Vaccine Effectiveness Among Health Workers in Azerbaijan
Acronym: VaccEffect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Public health and reforms Center of Ministry of Health (Other)
Collaborators: World Health Organization (Other); Ministry of Health of Azerbaijan Republic (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2-PHRC-2021
Record Dates: First submitted 2021-06-10; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-07

CONDITIONS: Vaccine Refusal; Covid19
MeSH Terms: conditions — Vaccination Refusal; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a prospective longitudinal cohort study, which will compare SARS-CoV-2 incidence among COVID-19 vaccinated and unvaccinated HWs who are eligible for COVID-19 vaccination in Azerbaijan.
  Upon approval of the protocol, all HWs working at six hospitals of Baku capital and who are eligible for COVID-19 vaccination will be offered to participate in the study and followed up regularly over time. The participation is completely voluntary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure group (Active Comparator): Healthcare workers vaccinated by any of the available COVID19 vaccine;
  Interventions: Biological: COVID-19 vaccine Observation of individuals who receive the COVID-19 vaccine
- Control group (Active Comparator): Have not received any doses of any form of COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccine Observation of individuals who receive the COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine Observation of individuals who receive the COVID-19 vaccine — To measure the effectiveness of COVID-19 vaccines against symptomatic laboratory-confirmed SARS-CoV-2 infection amongst hospital level health workers eligible for vaccination.

SUMMARY:
Many critical questions remain about the effectiveness of COVID-19 vaccines in real-world settings. These questions can only be answered in post-introduction vaccine effectiveness studies.

This protocol describes a prospective one-year cohort study of hospital-based HWs in Baku city of Azerbaijan to evaluate the effectiveness of COVID-19 vaccine in preventing laboratory-confirmed SARS-CoV-2 infection and COVID-19 disease. HWs are the target population in this study because HWs have been prioritized to be the first group to receive the vaccine in Azerbaijan and offer an early opportunity to evaluate the vaccine in a population in which it is critical that an effective vaccine be deployed.

HWs will be enrolled after the study protocol is approved by the local ethical review committee. All HWs eligible to be vaccinated with COVID-19 vaccine can be enrolled in the study, including those who intend to get vaccinated, those who don't plan on getting vaccinated, and those who are not sure. The target enrolment is 1500 HWs in six hospitals in Baku, the capital of Azerbaijan.

At enrolment, study participants will complete a baseline enrolment e-survey about demographics, clinical comorbidities, and work- and community-related behaviours related to infection risk. In addition, a baseline serology will be collected from participants at enrolment. No PCR testing for COVID19 virus will be done at the time of enrollment.

During the course of the study, participants will be actively followed for suspected symptomatic COVID-19 illness. Participants who meet a suspected case definition will be asked to have respiratory sample for SARS-CoV-2 by RT-PCR to be collected by trained HWs. PCR-positive samples from participants may also undergo genetic sequencing in or outside of Azerbaijan to identify the genetic makeup of the SARS-CoV-2 that caused the infection.

Finally, at 6 months and 12 months of the study, serology will be collected from participants to confirm and quantify the immunity after vaccination as a secondary objective. Serology will be tested for antibodies to SARS-CoV-2. Serology samples will be stored and may be sent to laboratories outside of Azerbaijan for advanced serologic testing.

Vaccine effectiveness should be analysed as described in the analysis section below.

In addition to the final analysis at the end of the one-year period, interim quarterly (every three months) analyses will be undertaken.

DETAILED DESCRIPTION:
2. Background and study rationale In late 2019 a novel severe acute respiratory syndrome - coronavirus 2 (SARS-CoV-2), which causes coronavirus disease 2019 (COVID-19), emerged. On January 30, 2020, WHO declared COVID-19 a public health emergency of international concern. On 11 March 2020, the World Health Organization declared COVID-19 a pandemic. The first case of COVID-19 was detected in Azerbaijan end of February, 2020, and since then 236,012 cases and 3,235 deaths has been reported in the country (data as of 8 March 2021).1

Effective and safe vaccines against COVID-19 are vital for controlling the pandemic. International collaborative efforts have accelerated the development of COVID-10 vaccines. As of 5 March 2021, there were 182 vaccines in pre-clinical development, and 79 vaccines in clinical development2. As of 18 February 2021, at least seven different vaccines across three platforms had been rolled out in countries, including the Coronac vaccine produced by Chinese company Sinopharm.

Evaluating the real-world COVID-19 vaccine performance is critical for understanding the risks and benefits of vaccination programs. Many factors impact real-world vaccine effectiveness (VE), including vaccine transportation and storage and how patients are vaccinated. In addition, the people who get the vaccine in clinical trials are often young and healthy, and therefore different from those who will receive vaccines in the real world. Post-licensing VE studies can also answer questions about effectiveness by age-group and underlying medical conditions, duration of vaccine protection, relative effectiveness of different vaccines, relative effectiveness of one dose vs. two doses, and effectiveness of the vaccine against new strains of SARS-CoV-2.

Health workers (HW) have been targeted for this study for a number of reasons. Azerbaijan has prioritized HWs for vaccination in line with the recommendations of the WHO SAGE and the European Technical Advisory Group on immunizations for use of COVID-19 vaccines when supply is limited. HWs provide a critical essential service in the COVID-19 pandemic response. HWs are at high risk of acquiring infection and associated morbidity and mortality, and also pose a risk of onward transmission to people who are also at high risk of serious COVID-19 outcomes. Ensuring that HWs receive an effective vaccine is also guided by the principle of reciprocity because HWs play critical roles in the COVID-19 response, working under intense and challenging conditions. Targeting HWs in this study offers an opportunity to determine the effectiveness of the vaccine in a population in which it is critical that an effective vaccine be deployed. While the HW population is not perfectly representative of the population of Azerbaijan, having an early understanding of the effectiveness of the vaccine in this population can inform decisions about vaccine use in the general population.

Immunization of HWs in Azerbaijan with Coronavac started in January 18, and the second dose has been administered to more than 60% of HWs by 15 March 2021. At the same time, it is estimated that 45-60% of health workers at the six target hospitals have received at least one dose and 60% of those have also received second dose of the vaccine.

Investigators propose to study the effectiveness of the COVID-19 vaccine in HWs in six selected hospitals in Baku city of Azerbaijan in order to answer critical questions about the real-world performance of COVID-19 vaccines in one of the key target groups for vaccination.

The stakeholders of this study include the following: Azerbaijan Republic Ministry of Health, The Public Health and Reforms Center of the Azerbaijan MOH, TABIB (which is subsidiary of Mandatory Health Insurance Agency of Azerbaijan that manages most hospitals in the country) health workers in the six hospitals and in Azerbaijan in general, the administration of the six study hospitals, and the World Health Organization.

2.1. Objectives 2.1.1. Primary objective To measure the effectiveness of COVID-19 vaccines against symptomatic laboratory-confirmed SARS-CoV-2 infection amongst hospital level health workers eligible for vaccination.

2.1.2. Secondary objectives

* What is the effectiveness of Covid-19 vaccine in preventing any laboratory- confirmed SARS-CoV-2 infection, including symptomatic and asymptomatic infection, as measured by infection detected by PCR and serology?
* How long does the COVID-19 vaccine confer protection against infection?
* What is vaccine effectiveness (VE) by age?
* What is VE by comorbidity?
* What is the VE in people who have been previously infected with SARS-CoV-2 compared with those who were previously uninfected?
* Does vaccine effectiveness vary by degree of exposure to COVID-19 patients in the hospital setting and physical distancing practices outside of the hospital?
* Does vaccine effectiveness vary by new strains of SARS-CoV-2 that may emerge?

  3. Methods 3.1. Study setting and population

The study will be conducted among health workers working in six hospitals in different districts of Baku, the capital of Azerbaijan republic. The number of employees in each hospital is provided in the Table below.

Hospitals in Baku are chosen for a number of reasons. The Baku capital is the largest city in the country with over 3 million inhabitants. It has the largest hospitals in the country and the largest number of hospital-based HWs of any city in the country. Baku has been and still is at the forefront of fight with pandemic; the largest number of infections have occurred in Baku, and the largest number of COVID-19 patients requiring medical care are being treated in Baku hospitals. In addition, conducting the study in Baku will facilitate issues related to monitoring, supervision and logistics,. given the nation-wide quarantine-related restrictions and limitations to regional travel. Investigators selected a convenience samples of hospitals in various parts of Baku city.

The study population will be composed of HWs in the above hospitals, eligible for vaccination, with no contraindication to receive COVID-19 vaccine. HWs include all categories of staff working in these hospitals, including clinical and non-clinical/administrative staff and staff with direct patient interaction and those without direct patient interaction.

All HWs who are eligible for vaccination, according to MoH guidelines, will be offered enrolment, regardless of their intention to receive the COVID-19 vaccine. Currently, all HWs are eligible to receive vaccines unless they have contraindications, such as severe allergic reactions to previous vaccinations. Along with HWs, the educators, police and military personnel as well as all citizens >50 years of age are eligible to receive vaccines unless there are contraindications including allergies to vaccine incipient/excipients or previously confirmed allergic reaction to vaccination or current viral or bacterial infections.

This study will ensure follow up of enrolled participants via serology, respiratory swabs, and questionnaires. Participants may receive COVID19 vaccine during the study period but not as part of this study.

Efforts will be made to enroll all HW as close as possible to the time of their first vaccination.

Study staff will coordinate with hospital administration in order to ensure that the study will not interfere with vaccine administration.

ELIGIBILITY:
Study Population The study population will be composed of health workers in the selected 7 hospitals, eligible for vaccination, with no contraindication to receive COVID-19 vaccine. Health Workers include all categories of staff working in the hospitals, including clinical and non-clinical/administrative staff and staff with direct patient interaction and those without direct patient interaction.

Criteria

Inclusion Criteria:

- All Health Workers in selected 7 hospitals eligible to receive the COVID-19 vaccination.

Exclusion Criteria:

* Health Workers who are not eligible for COVID-19 vaccination or have a contraindication to vaccination.
* Health Workers who do not work at selected 7 hospitals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine effectiveness | 12 months
  Weekly symptom questionnaire for all symptomatic vaccinated participants will identify potential new SARS-CoV-2 infection among vaccinated participants.
Post-vaccination COVID-19 cases | 12 months
  COVID-19 PCR testing for all symptomatic vaccinated participants will identify new SARS-CoV-2 infection among vaccinated participants.

SECONDARY OUTCOMES:
Vaccine effectiveness by age | 12 months
  The enrollment questionnaire includes age of each participant. Data will be stratified by age at the time of analysis.
Vaccine effectiveness in participants with various co-morbidities | 12 months
  The enrollment questionnaire will assess the existence of specific co-morbidities among participants, including (but not limited to) heart disease, autoimmune disease, chronic liver disease and chronic kidney disease. Data will be stratified by co-morbidity at the time of analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health and Reforms Center of Ministry of Health, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.isim.az
- See also: Related Info — http://www.ejcs.org
- Available data/document: Study Protocol — http://www.isim.az